CLINICAL TRIAL: NCT05455476
Title: Telehealth CBT to Address Social Isolation in Veterans With Chronic Pain
Brief Title: Pain and Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4091-P
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain
Keywords: Loneliness; Chronic pain; social isolation; social connection
MeSH Terms: conditions — Chronic Pain; Social Isolation

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two interventions.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcomes assessors will not know what condition that the participant was allocated to, nor will the statistician who is one of the co-investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT for Loneliness (Experimental): CBT delivered over the course of 8, ~45 minute sessions delivered via telehealth more centrally focused addressing factors contributing to loneliness and social isolation.
  Interventions: Behavioral: CBT for Loneliness
- CBT for Chronic Pain (Active Comparator): CBT delivered over the course of 8, ~45 minute sessions delivered via telehealth broadly focused on increasing quality of life despite being in pain.
  Interventions: Behavioral: CBT for Chronic Pain

INTERVENTIONS:
Behavioral: CBT for Loneliness — CBT delivered over the course of 8, ~45 minute sessions delivered via telehealth more centrally focused addressing factors contributing to loneliness and social isolation.
  Arms: CBT for Loneliness
Behavioral: CBT for Chronic Pain — CBT delivered over the course of 8, ~45 minute sessions delivered via telehealth broadly focused on increasing quality of life despite being in pain.
  Arms: CBT for Chronic Pain

SUMMARY:
Loneliness-feeling socially isolated-is a stressor that is associated with chronic pain. The investigators will first conduct a small trial of Cognitive Behavioral Therapy for Loneliness (CBT-L)in Veterans with chronic pain reporting loneliness. After completing this small trial, the investigators will randomize-like a flip of a coin-a total of 40 participants to receive either CBT-L or CBT for Chronic Pain. The investigators will assess loneliness, the quality and quantity of social interactions, and pain outcomes such as pain-related interference, and thinking the worst about one's pain at baseline and after the treatment period. The investigators will also track participant flow, therapist adherence to the manual, participant homework completion, and participant satisfaction with the treatment.

DETAILED DESCRIPTION:
Loneliness-a subjective emotional state characterized by the perception of social isolation-is a psychosocial stressor that is associated with increased mortality and chronic pain. Individuals who have chronic pain and report loneliness experience greater pain-related interference in activities, depression, and suicidal ideation. Importantly, there are potentially effective interventions that can be used to decrease loneliness; however, there are no studies that have directly intervened on loneliness among Veterans with chronic pain. Cognitive-Behavioral Therapy for Loneliness (CBT-L) intervenes on loneliness by addressing negative beliefs that perpetuate loneliness, increase negative affect, and reduce one's ability to engage in social activities. For a Veteran with chronic pain, this is critical as addressing negative affect, and having a sense that one has social support and engages social support are key aspects of increasing functioning. While CBT for Chronic Pain (CBT-CP) comprises skills to promote social functioning, more robust efforts may be needed to better address lonely while also addressing functional impairment.

The proposed two-year study uses a novel application of a brief, phone-delivered, evidence-based intervention, CBT-L, to decrease loneliness by modifying socially-relevant maladaptive thinking patterns, increasing engagement in enjoyable and social activities, and improving problem solving skills. Participants will be recruited nationally using online advertising. The objectives of the current proposal are to adapt CBT-L to optimize its impact on Veterans with chronic pain, examine if the recruitment, retention, and treatment delivery is feasible and if CBT-L is acceptable to participants, and assess parameters of key outcomes among participants randomized to receive CBT-L versus CBT-CP to inform a subsequent larger clinical trial.

To achieve these objectives, the investigators will adapt a manual through an evidence-based, iterative process then conduct one-arm trial of CBT-L (n=8) in Veterans with chronic pain reporting loneliness. After refining the manual and procedures following the one-arm trial, the investigators will randomize a total of 40 participants to receive either CBT-L or CBT-CP. The investigators will assess loneliness, the quality and quantity of social interactions, and pain outcomes such as pain-related interference, and pain catastrophizing at baseline and after the treatment period. The investigators will also track participant flow, therapist adherence to the manual, participant homework completion and participant satisfaction with the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Are English-speaking
* Are 18 years of age or older
* Have access to a phone or computer
* Report pain that occurs on at least half the days for six months or more
* Score at least 4 (of 10) on each of the three items on the PEG (Pain intensity, and Pain interference in Enjoying activities and General activities)
* Screen positive for loneliness by scoring at least a T-score > 60 on the NIH Toolbox loneliness scale

Exclusion Criteria:

* Do not understand informed consent
* Had a recent or have an upcoming surgery
* Have significant unstable or uncontrolled medical conditions, including cancer requiring ongoing oncology treatment
* Active severe substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisham Ashrafioun, PhD, Principal Investigator — VA Finger Lakes Healthcare System, Canandaigua, NY
Locations (1):
- VA Finger Lakes Healthcare System, Canandaigua, NY, Canandaigua, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were recruited through a case finding procedure of VHA medical records.
Pre-assignment Details: The first 8 participants all received CBT for Loneliness after a baseline assessments. For the next 40 participants, participants in both conditions receive a baseline assessment and then were randomized to either CBT for Chronic Pain or CBT for Loneliness.
Period: Overall Study
Arm/Group | CBT for Loneliness | CBT for Chronic Pain
Started | 28 | 20
Completed | 18 | 13
Not Completed | 10 | 7

BASELINE CHARACTERISTICS:
Population: Two participants in the CBT for Loneliness arm were consented, but did not complete the baseline assessment. The other participant withdrew.
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT for Loneliness | CBT for Chronic Pain | Total
Number analyzed (Participants) | 25 | 20 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (10.7) | 52.8 (14.3) | 53.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 20 | 16 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 21 | 20 | 41
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 5 | 11
  White | 16 | 11 | 27
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
UCLA Loneliness Scale [Mean (Standard Deviation); unit: units on a scale] — The scores range from 20-80 with higher scores indicating worse outcome.
  units on a scale | 56.0 (10.4) | 56.8 (10.3) | 56.4 (10.2)
Brief Pain Inventory-Pain Interference [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 70 with higher scores indicating worse outcomes.
  units on a scale | 52.5 (13.2) | 55.4 (8.9) | 53.8 (11.3)
Tampa Scale of Kinesiophobia [Mean (Standard Deviation); unit: units on a scale] — Scores range from 17 to 68 with higher scores indicating worse outcomes.
  units on a scale | 45.8 (7.9) | 46.3 (7.9) | 46.0 (7.7)
PROMIS Depression [Mean (Standard Deviation); unit: units on a scale] — The scores range from 4-20 with higher scores indicating worse outcome.
  units on a scale | 10.8 (4.3) | 13.1 (3.6) | 11.8 (4.1)
PROMIS Anxiety [Mean (Standard Deviation); unit: units on a scale] — The scores range from 4-20 with higher scores indicating worse outcome.
  units on a scale | 10.9 (4.1) | 13.0 (3.0) | 11.8 (3.7)
Pain Catastrophizing Scale [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0 to 52 with higher scores indicating worse outcomes.
  units on a scale | 31.9 (11.5) | 30.2 (9.0) | 31.2 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Loneliness
Description: Loneliness will be measured using the UCLA Loneliness Scale. A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item as 1 (never), 2 (rarely), 3 (sometimes) or 4 (often). The scores range from 20-80 with higher scores indicating worse outcome.
Time Frame: baseline to 1-month post-treatment
Population: Participant flow includes participants from the one-arm trial. Participants reported in the outcomes do not include participants from the one-arm trial because there was not a one-month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT for Loneliness | CBT for Chronic Pain
Number analyzed (Participants) | 12 | 13
score on a scale | -6.6 (7.2) | -2.5 (9.1)

2. Primary Outcome: Mean Change in Pain Interference
Description: Pain interference will be measured using the Brief Pain Inventory Pain Interference subscale. The pain interference subscale comprises 7 items assessing the extent to which pain interferes with various aspects of one's life (e.g., mood, sleep, daily activities) with scores ranging from 0 to 70. Higher scores represent greater pain-related interference in activity.
Time Frame: baseline to 1-month post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score of a scale
Arm/Group | CBT for Loneliness | CBT for Chronic Pain
Number analyzed (Participants) | 11 | 12
score of a scale | -2.4 (2.5) | -0.5 (1.6)

3. Secondary Outcome: Mean Change in Social Interactions
Description: Duke Social Support Index assesses several domains of perceived social support, including social network size, social interaction, social satisfaction, and instrumental social support. Higher scores indicate a higher quality of social interactions. Scores range from 0 to 37.
Time Frame: baseline to 1-month post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | CBT for Loneliness | CBT for Chronic Pain
Number analyzed (Participants) | 12 | 13
score on scale | -0.33 (2.5) | 0.46 (2.5)

4. Secondary Outcome: Mean Change in Fear of Pain
Description: Fear of movement due to pain will be measured using the Tampa Scale of Kinesiophobia. The scores range from 17-68 with higher scores indicating worse outcome.
Time Frame: baseline to 1-month post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT for Loneliness | CBT for Chronic Pain
Number analyzed (Participants) | 12 | 13
score on a scale | -3.17 (6.0) | -0.54 (5.9)

5. Other Pre Specified Outcome: Mean Change in Depression
Description: Depression will be measured using the PROMIS tool. The scores range from 4-20 with higher scores indicating worse outcome.
Time Frame: baseline to 1-month post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT for Loneliness | CBT for Chronic Pain
Number analyzed (Participants) | 12 | 13
score on a scale | -3.25 (4.1) | -0.3 (4.1)

6. Other Pre Specified Outcome: Mean Change in Anxiety
Description: Anxiety will be measured using the PROMIS tool. The scores range from 4-20 with higher scores indicating worse outcome.
Time Frame: baseline to 1-month post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT for Loneliness | CBT for Chronic Pain
Number analyzed (Participants) | 12 | 13
score on a scale | -3.7 (3.8) | -0.6 (3.9)

7. Other Pre Specified Outcome: Mean Change in Pain Catastrophizing
Description: The Pain Catastrophizing Scale (PCS) is a 13-item measure, with each item rated on a 5-point rating scale (0 = "Not at all" to 4 = "All the time"). The measure is divided into three subscales: magnification, rumination, and helplessness. Scores range from 0 to 52 with higher scores indicate greater pain catastrophizing.
Time Frame: baseline to 1-month post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT for Loneliness | CBT for Chronic Pain
Number analyzed (Participants) | 12 | 13
score on a scale | -7.1 (10.1) | -2.3 (12.4)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up (baseline assessment, post-treatment assessment, 1-month follow-up; 8 intervention session; ~3 months)
Arm/Group | CBT for Loneliness | CBT for Chronic Pain
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/20
Serious Adverse Events (participants affected / at risk) | 3/28 | 2/20
Other Adverse Events (participants affected / at risk) | 7/28 | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CBT for Loneliness (N=28) | CBT for Chronic Pain (N=20)
Hospital admission - COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — unrelated to study
Hospital admission - falls (Nervous system disorders) | 1 | 0 — unrelated to study
Hospital admission - Nerve pain (Nervous system disorders) | 1 | 0
Hospital admission - suicidal ideation (Psychiatric disorders) | 0 | 1 — unrelated to study
Hospital admission - hypokalemia (Metabolism and nutrition disorders) | 0 | 1 — unrelated to study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CBT for Loneliness (N=28) | CBT for Chronic Pain (N=20)
Emergency department visit - pain (Musculoskeletal and connective tissue disorders) | 1 | 1 — unrelated to study
Emergency department visit - head pain (Nervous system disorders) | 0 | 2 — unrelated to study
Emergency department visit - nausea, chest pain (Gastrointestinal disorders) | 0 | 1 — unrelated to study
Psychological distress (Social circumstances) | 3 | 2 — unrelated to study
Emergency department visit - pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — unrelated to study
Emergency department - fall (Nervous system disorders) | 2 | 0 — unrelated to study
Emergency department visit - erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 — unrelated to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT05455476/Prot_SAP_001.pdf
  • Informed Consent Form (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT05455476/ICF_000.pdf